CLINICAL TRIAL: NCT02803437
Title: Drug Use Investigation of Xofigo, Castration Resistant Prostate Cancer With Bone Metastases
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18212
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: Castration-resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Xofigo / Cohort 1: Patients suffered from CRPC with bone metastases are enrolled after the physician's decision of Xofigo treatment under the routine clinical practice.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY 88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY 88-8223) — Xofigo treatment will be performed according to the product label in Japan under the routine clinical practice.

SUMMARY:
This study is a Japanese post-marketing surveillance (PMS) which is required by the regulatory authorities. General objective of PMS is to confirm the clinical usefulness, especially the safety profile of a drug under the routine clinical practice.

DETAILED DESCRIPTION:
This is a local, non-interventional, multi-center, single-cohort study using primary data of patients treated with Xofigo for the indication of castration resistant prostate cancer (CRPC) with bone metastases. A total of 300 patients (valid for safety analysis) are enrolled within 18 months.

During the observation period (i.e. up to 6 months), safety and effectiveness information is collected. Since patient's visit occurs under the routine clinical practice, the study protocol does not define exact referral dates for those visits. The physician records patient data as defined in the protocol.

The extended follow-up period is to collect bone fractures and survival with post-treatment information after Xofigo under the real-world in Japan.

The results of this study (except of extended follow-up period) have to be submitted to the Japanese regulatory authorities as a part of the reexamination period (8 years). This study is conducted in accordance with Article 14-4 (re-examination) of the Pharmaceutical Affairs Law, and Good Post-marketing Surveillance Practice from a ministerial ordinance of Ministry of Health, Labor and Welfare in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffered from CRPC with bone metastases
* Patients for whom the decision to initiate treatment with Xofigo is made as per physician's routine clinical practice.
* Xofigo treatment naïve

Exclusion Criteria:

* Patients treated Xofigo previously
* Patients participating in an investigational program with interventions outside of routine clinical practice

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffered from castration resistant prostate cancer with bone metastases
Sampling Method: Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Number of adverse events as a measure of safety | Up to 6 months
  Events will be summarized by frequency tables (e.g. absolute and relative frequencies) using the MedDRA coding system
Number of adverse drug reactions as a measure of safety | Up to 6 months
  Events will be summarized by frequency tables (e.g. absolute and relative frequencies) using the MedDRA coding system

SECONDARY OUTCOMES:
Change in laboratory findings (e.g. ALP, bone markers) | From Baseline up to 6 month
Change in analgesic use as a surrogate of pain status | From Baseline up to 6 month
Number of patients with bone fractures | Up to 3 years
Survival rate | Up to 3 years
Post-treatment information | Up to 3 years
  Comprises information of post-treatment medication/ therapy for prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Result] Hosono M, Uemura H, Kakehi Y, Masumori N, Takahashi S, Okayama Y, Sunaya T, Horio T, Kinuya S. [Exploratory Analysis Results from Post-marketing Surveillance Study of Radium-223 in Japanese Patients with Castration-resistant Prostate Cancer and Bone Metastases: Subgroup Analysis by Age]. Kaku Igaku. 2021;58(1):91-101. doi: 10.18893/kakuigaku.oa.2105. Japanese. PMID 34645727
- [Result] Uemura H, Masumori N, Takahashi S, Hosono M, Kinuya S, Sunaya T, Horio T, Okayama Y, Kakehi Y. Real-world safety and effectiveness of radium-223 in Japanese patients with castration-resistant prostate cancer (CRPC) and bone metastasis: exploratory analysis, based on the results of post-marketing surveillance, according to prior chemotherapy status and in patients without concomitant use of second-generation androgen-receptor axis-targeted agents. Int J Clin Oncol. 2021 Apr;26(4):753-763. doi: 10.1007/s10147-020-01850-3. Epub 2021 Feb 11. PMID 33575828
- [Result] Masumori N, Kakehi Y, Hosono M, Kinuya S, Takahashi S, Okayama Y, Sunaya T, Horio T, Uemura H (2020) Post-marketing Surveillance （PMS） Study for Safety and Effectiveness of Radium-223 in Japanese Patients with CRPC and Bone Metastases in Real-world Settings: Exploratory Analysis on Treatment Completion of Six Cycles of Radium-223 and Discontinuation. Medical Consultation & New Remedies 57:705-717
- [Result] Takahashi S, Uemura H, Masumori N, Kinuya S, Hosono M, Okayama Y, Sunaya T, Horio T, Kakehi Y (2020) Safety and effectiveness of radium-223 in Japanese patients with CRPC and bone metastases in real world-settings: The results of post-marketing surveillance (PMS). Japanese Journal of Urological Surgery 33(4):435-449